CLINICAL TRIAL: NCT05008263
Title: Competitive Accuracy of Radiological Imaging Compared to Liver Biopsy in Patients With Liver Fibrosis
Status: Completed | Type: Observational
Sponsor: Vilnius University (Other)
Responsible Party: Sponsor
Other Study IDs: 158200-18/7-1053-552
Record Dates: First submitted 2021-06-23; First posted 2021-08-17 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-06

CONDITIONS: Liver Fibroses; Liver Cirrhosis
Keywords: Liver fibrosis; Liver cirrhosis; Liver biopsy; Shear wave imaging; Dynamic liver scintigraphy
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with viral chronic liver disease at primary diagnosis: Patients with primary diagnosis of viral hepatitis B and hepatitis C who was referred for liver biopsy. All patients underwent liver shear wave elastography and dynamic liver scintigraphy evaluating liver physical and functional changes shortly prior to liver biopsy procedure.
  Interventions: Diagnostic Test: Liver elastography (2D-SWE); Diagnostic Test: Liver scintigraphy with 99mTc-mebrofenin

INTERVENTIONS:
Diagnostic Test: Liver elastography (2D-SWE) — All patients were referred for 2D-SWE liver elastography and liver liver scintigraphy with 99mTc-mebrofenin prior to liver biopsy.
Diagnostic Test: Liver scintigraphy with 99mTc-mebrofenin — All patients were referred for 2D-SWE liver elastography and liver liver scintigraphy with 99mTc-mebrofenin prior to liver biopsy.

SUMMARY:
The study "Competitive Accuracy of Radiological Imaging Compared to Liver Biopsy in Patients With Liver Fibrosis" is designed to test the accuracy of non-interventional radiological imaging and compare its results with the "gold standard" liver biopsy. This is prospective non-randomized single patient group study.

ELIGIBILITY:
Inclusion Criteria:

* chronic liver disease
* signed informed consent
* liver biopsy indicated by treating gastroenterologist/infectologist

Exclusion Criteria:

* non-corrected blood coagulation tests
* acute liver disease
* age below 18 years or above 80 years
* disagreement to participate in the study
* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary diagnosis of chronic viral liver disease who are referred treating gastroenterologist/infectologist for liver biopsy prior to treatment.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Ultrasound elastography comparison to histological examination of liver biopsy specimen | Baseline only
  Liver stiffness measured by ultrasound elastography (2D-SWE) in kPa is compared to histological examination of liver biopsy specimen at a single time point before initiating antiviral treatment.
Dynamic liver scintigraphy with 99mTc-mebrofenin comparison to histological examination of liver biopsy specimen I | Baseline only
  Dynamic liver scintigraphy with 99mTc-mebrofenin parameter liver clearance (%/min/m2) is compared to histological examination of liver biopsy specimen at a single time point before initiating antiviral treatment.
Dynamic liver scintigraphy with 99mTc-mebrofenin comparison to histological examination of liver biopsy specimen II | Baseline only
  Dynamic liver scintigraphy with 99mTc-mebrofenin parameter uptake time (min.) is compared to histological examination of liver biopsy specimen at a single time point before initiating antiviral treatment.
Dynamic liver scintigraphy with 99mTc-mebrofenin comparison to histological examination of liver biopsy specimen III | Baseline only
  Dynamic liver scintigraphy with 99mTc-mebrofenin parameter liver excretion (30 min./peak ratio) is compared to histological examination of liver biopsy specimen at a single time point before initiating antiviral treatment.

SECONDARY OUTCOMES:
Comparison of radiological imaging tests between each other I | Baseline only
  Liver stiffness measured by ultrasound elastography (2D-SWE) in kPa is compared to liver clearance measured by dynamic liver scintigraphy with 99mTc-mebrofenin.
Comparison of radiological imaging tests between each other II | Baseline only
  Liver stiffness measured by ultrasound elastography (2D-SWE) in kPa is compared to tracer excretion measured by dynamic liver scintigraphy with 99mTc-mebrofenin.
Comparison of radiological imaging tests between each other III | Baseline only
  Liver stiffness measured by ultrasound elastography (2D-SWE) in kPa is compared to tracer uptake time measured by dynamic liver scintigraphy with 99mTc-mebrofenin.

CONTACTS AND LOCATIONS:
Overall Officials: Algirdas E Tamosiunas, MD, PhD, Principal Investigator — Vilnius University
Locations (1):
- Vilnius University, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: Undecided